CLINICAL TRIAL: NCT04898400
Title: Role of Eosinophils in Human Adipose Tissue Metabolism
Brief Title: Eosinophils in Human Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elena Anna (Eleanna) De Filippis, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-000959
Record Dates: First submitted 2021-05-16; First posted 2021-05-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with Obesity (Experimental): Subjects will be recruited to undergo endoscopic sleeve gastroplasty. The subjects will be studied at baseline, 30, 60, 90 days after procedure
  Interventions: Procedure: endoscopy sleeve gastroplasty

INTERVENTIONS:
Procedure: endoscopy sleeve gastroplasty — endoscopic procedure for weight loss

SUMMARY:
The purpose of this study is to better understand the interactions between the innate immune system, in particular eosinophils (EOS), and adipose tissue (AT) in human health and in disease states such as obesity and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI>30 kg/m2).
* Evidence of insulin resistance as defined by hemoglobin A1c > 5.7%.
* Mayo Clinic patients evaluated by Dr. Rahul Pannala.
* Pursue an endoscopic gastroplasty at Mayo Clinic Arizona in the Gastroenterology department.
* Equal distribution of gender.
* 18 yo older of age.
* BMI>30 kg/m2.
* Nonsmoker.
* Taking no medication affecting glucose or lipid metabolism.
* No more than 5% change in body weight in the previous 6 months.
* Mostly sedentary (engaging in strenuous exercise (> 70% max HR) less than 3 times a week).
* Not be receiving corticosteroid therapy.
* Have no history of asthma, COPD or atopic syndrome, or autoimmune disease (Ulcerative colitis, Chron's disease, eosinophilic esophagitis, any rheumatologic disease such as lupus, rheumatoid arthritis, Sjogren syndrome).

Exclusion Criteria:

* <17 years of age.
* BMI <30 kg/m2.
* Smoker.
* Taking medication affecting glucose or lipid metabolism.
* Greater than 5% change in body weight within the previous six months.
* Engage in strenuous exercise (>70% max HR) less than 3 times a week.
* Receiving corticosteroid therapy.
* Have a history of asthma.
* History of COPD or atopic syndrome.
* History of autoimmune disease (Ulcerative colitis, Chron's disease, eosinophilic esophagitis, any rheumatologic disease such as lupus, rheumatoid arthritis, Sjogren syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
weight loss | at 30 days post-intervention
  total body weight
weight loss | at 60 days post-intervention
  total body weight
weight loss | at 90 days post-intervention
  total body weight
fat mass | at 30 days post-intervention
  % fat mass will be estimated by bioimpedence
fat mass | at 60 days post-intervention
  % fat mass will be estimated by bioimpedence
fat mass | at 90 days post-intervention
  % fat mass will be estimated by bioimpedence
AT-EOS content | at baseline
  subcutaneous fat biopsy will be processed to extract stromal vascular fraction (SVF) which will contain eosinophils. The SVF will be run trough flow cytometry to get an estimated count to be reported as a ratio over the total number of cells
AT-EOS content | at 90 days post-intervention
  subcutaneous fat biopsy will be processed to extract stromal vascular fraction (SVF) which will contain eosinophils. The SVF will be run trough flow cytometry to get an estimated count to be reported as a ratio over the total number of cells

SECONDARY OUTCOMES:
insulin sensitivity | at baseline and 90 days post-intervention
  mixed meal test
inflammation | at 30 days post-intervention
  Plasma will be isolated during fasting condition. MCP-1, TNFa, IL-4, IL-13, Leptin, adiponectin will be assessed via Multiplex ELISA
inflammation | at 60 days post-intervention
  Plasma will be isolated during fasting condition. MCP-1, TNFa, IL-4, IL-13, Leptin, adiponectin will be assessed via Multiplex ELISA
inflammation | at 90 days post-intervention
  Plasma will be isolated during fasting condition. MCP-1, TNFa, IL-4, IL-13, Leptin, adiponectin will be assessed via Multiplex ELISA
adipose tissue inflammation | at baseline
  subcutaneous fat biopsy will be processed to obtain mRNA. mRNA levels for MCP-1, TNFa, IL-4, IL-13, Leptin, adiponectin gene will be assessed via qPCR
adipose tissue inflammation | at 90 days post-intervention
  subcutaneous fat biopsy will be processed to obtain mRNA. mRNA levels for MCP-1, TNFa, IL-4, IL-13, Leptin, adiponectin gene will be assessed via qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Elena Anna O. De Filippis, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States